CLINICAL TRIAL: NCT06266936
Title: Smart Life Smart Living Intercontinental - Medical Students' Cohort
Acronym: SL2i-MSC
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Other Study IDs: EssaiClinique_SL2i-MSC
Record Dates: First submitted 2023-12-22; First posted 2024-02-20 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Mental Health Issue; Student Burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort with health students
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — The study involves longitudinal monitoring of the state of health of the specific population of students in care courses, from their entry into university studies (first year) until their final year of study, i.e. from 5 to 13 years depending on the course and the different universities.

SUMMARY:
The question of the well-being, quality of life and mental health of care students is unanimously considered to be a central issue among young adults. According to the French Ministry of Higher Education and Research, there will be 194,752 care students in France in 2021-2022. The quality of life and well-being of health students can be affected at several levels. The first is mental health. In France, the mental health of these students has deteriorated considerably in recent years. According to a 2017 survey of 21,768 French medical students, 66% of them had an anxiety disorder and 27% a depressive syndrome. In addition, a number of risk factors have been identified for the mental health of health students.

The aim of the study is to carry out a longitudinal evaluation of the mental health status of care students during their university studies in France through anxiety, depression and perceived stress.

ELIGIBILITY:
Inclusion Criteria:

* students who are regularly enrolled in healthcare courses at a French university

Exclusion Criteria:

* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study concerns students over the age of 18 who are regularly enrolled in healthcare courses at a French university.
  The study involves longitudinal monitoring of the state of health of the specific population of students in care courses, from their entry into university studies (first year) until their final year of study, i.e. from 5 to 13 years depending on the course and the different universities.
Sampling Method: Non-Probability Sample
Enrollment: 1564 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2044-09 (Estimated); Study Completion 2044-12 (Estimated)

PRIMARY OUTCOMES:
Synthetic score on standardized assessment scale of anxiety | 1 hour
  State Trait Anxiety Inventory (STAI)

SECONDARY OUTCOMES:
Synthetic score on standardized assessment scale of mental health | 1 hour
  Hospital Anxiety Depression (HAD)
Synthetic score on standardized assessment scale of stress | 1 hour
  Scale and Perceived Stress Scale (PSS-14)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Vuillerme, PhD, Study Chair — University Grenoble Alps

IPD SHARING:
Plan to Share IPD: Undecided